CLINICAL TRIAL: NCT02151721
Title: Phase I of Vorinostat-Iressa Combined Therapy on Resistance by BIM Polymorphysim in EGFR Mutant Lung Cancer
Acronym: VICTORY-J
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kanazawa University (Other)
Responsible Party: Principal Investigator, Seiji Yano, M.D., Ph.D., Chairman, Division of Medical Oncology Cancer Research Institute, Kanazawa University., Kanazawa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H25-S-I-005
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Vorinostat; Gefitinib; BIM polymorphism; EGFR-TKI resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vorinostat, gefitinib, combination (Experimental): single arm vorinostat plus gefitinib
  Interventions: Drug: Vorinostat, gefitinib

INTERVENTIONS:
Drug: Vorinostat, gefitinib — Vorinostat 200, 300, or 400 mg orally once daily on days 1-7 with washout on days 8-14 plus gefitinib 250 mg orally once daily on days 1-14
  Other Names: Zolinza; Iressa

SUMMARY:
* Gefitinib is an orally active epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI). However, 20-30% of patients with EGFR-activating mutations show intrinsic resistance to EGFR-TKI.
* EGFR-mutant non-small cell lung cancer (NSCLC) cells with BIM (BCL2L11) deletion polymorphism show the impaired generation of BIM with the proapoptotic BH3 domain, as well as resistance to EGFR-TKI-induced apoptosis.
* Both BIM polymorphism (12.9%) and EGFR mutations (50% in lung adenocarcinoma) are more prevalent in the East Asian than in Caucasian populations. BIM is a BH3-only proapoptotic member of the Bcl-2 protein family. BIM upregulation is required for apoptosis induction by EGFR-TKI in EGFR-mutant NSCLC.
* Vorinostat (suberoylanilide hydroxamic acid [SAHA]) is a small-molecule inhibitor of histone deacetylase (HDAC) and induces cell differentiation, cell cycle arrest, and apoptosis in several tumor cells. HDAC inhibition can epigenetically restore BIM function and death sensitivity of EGFR-TKI in patients with EGFR-mutant NSCLC in whom resistance to EGFR-TKI is associated with a common BIM polymorphism. EGFR-TKI resistance due to the BIM polymorphism may be able to be circumvented in combination with HDAC inhibition of vorinostat with gefitinib in NSCLC.

DETAILED DESCRIPTION:
* A cohort of three patients will be treated at each dose level for one cycle (28 days per cycle).
* Treatment will be continued if no DLTs are recorded, and three patients will be treated at the next higher dose level.
* If a patient of the cohort develops a DLT, however, another cohort of three patients will be treated for 1 cycle.
* If more DLTs do not develop, dose escalation continues.
* If more than one of three patients develop a DLT at any dose level, another cohort of three patients will be treated at the next lower dose level.
* If no DLTs are recorded in any of the cohorts, the number of patients per cohort will be increased from 3 to 6.
* Up to 12 patients will be enrolled at the MTD.
* Therefore, the phase II dose for this combined therapy will be defined as the highest dose level at which six patients were treated and less than three DLTs developed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed NSCLC (excluding squamous cell carcinoma)
* NSCLC of clinicopathologic stage IIIB or IV for which radical radiation therapy is impracticable, or recurrence after surgery
* EGFR mutations (deletion of exon 19 and L858R mutation of exon 21) for which the clinical benefits of an EGFR-TKI (gefitinib or erlotinib) are recognized by testing methods that are listed by the national health insurance
* Having a history of treatment with an EGFR-TKI (gefitinib or erlotinib) and a history of pathology deterioration during treatment
* Having a history of treatment with cytotoxic anticancer agents (not including pre- or postoperative chemotherapy that has passed 1 or more year from the day of final administration)
* Confirmed BIM polymorphism by the PCR fragment analytical method and the sequence method at the central laboratory
* Having a lesion measureable according to the RECIST guidelines revised version 1.1 (20 mm or larger in 10-mm slice CT, 10 mm or larger in 5-mm slice CT, 15 mm or larger in the minor axis of a lymph node). Confirmed advance of the pathology at the site of irradiation after irradiation in a patient who only has an irradiated lesion
* Ages 20 years and older
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1 at the time of consent acquisition
* Having adequate bone marrow (neutrophil count: 1,500/L, Platelet count: 100,000/L), hepatic (total bilirubin level: 1.5-fold or less of the upper limit of reference value at each institution), renal (creatinine level: 1.5 mg/dL), and respiratory functions (PaO2: 70 torr or SpO2: 94%) within 14 days before entry.
* An estimated life expectancy of 12 or more weeks after the onset of protocol treatment
* A patient whose acute toxicities of prior treatments have recovered to the baseline level in the most recent prior treatment, excepting adverse events considered not to be of safety concern at the discretion of the investigator (subinvestigator)
* A patient negative for the urinary pregnancy test to be performed at the time of screening prior to the onset of protocol treatment
* Acquisition of written informed consent to participate in the present study from the patient after receiving a satisfactory explanation about study details

Exclusion Criteria:

* Within 4 weeks after the final administration of a cytotoxic anticancer agent. Allowable enrollment when a 7-day washout is completed after the final administration of an EGFR-TKI. Surgery of a primary tumor or to the mediastinum must be completed at least 6 months before the onset of protocol treatment.
* Radiotherapy to the lungs considered necessary at the time of study entry or in the near future.
* Having an interstitial lung disease (including acute pulmonary disorder, interstitial pneumonia, and drug inducibility) or having a history thereof.
* Having radiation pneumonitis or having a history thereof.
* Having a large volume of or uncontrollable pleural effusion, ascites, or pericardial effusion
* Detection of known EGFR-TKI resistance acquired by mutations of the genes, e.g., T790M.
* Having a serious infection and other serious complications (e.g., gastrointestinal bleeding).
* Suffering from a severe or poorly controlled systemic disease (e.g., unstable or decompensated respiratory disease, heart disease, renal disease, and liver disease)
* Having an active, as well as poorly controlled or symptomatic metastasis to the central nervous system (involving cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, or invasion due to disease progress). Even with a history of metastasis to the central nervous system or of spinal compression.
* Having an active double cancer.
* Verified HBs antigen positivity or HCV antibody positivity (excluding the case of confirmed HCV-RNA negativity)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-02-20 (Estimated); Study Completion 2018-02-20 (Estimated)

PRIMARY OUTCOMES:
MTD (Maximum Tolerated Dose) | Second cycle (Day 28)
  MTD (Maximum Tolerated Dose)defined as the highest dose level at which < 2 out of 6 patients experienced a DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Seiji Yano, MD, PhD, Principal Investigator — Kanazawa University Hospital
Locations (5):
- Japan (5):
  - Nagoya University Graduate School of Medicine, Nagoya, Aichi-ken
  - Institute of Biomedical Research and Innovation Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
The 12th patient in stage 3 was registered.